CLINICAL TRIAL: NCT01531816
Title: Early Rehabilitation in Critically Ill Children, a Pilot Study
Brief Title: Early Rehabilitation in Critically Ill Children Pilot Study
Acronym: WeeHab in PCCU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-008
Record Dates: First submitted 2012-02-07; First posted 2012-02-13 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Critical Illness
Keywords: Pediatrics,; Critically ill Children; immobility
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm: Study Intervention (Experimental): Cycle ergometry and/or Interactive video-game
  Interventions: Device: Early Rehabilitation intervention

INTERVENTIONS:
Device: Early Rehabilitation intervention — 1. Passive mobility: cycle ergometer
  2. Active mobility: interactive video-game (X Box 360 Kinect) Each intervention will be applied for a maximum of 2 days respectively. If a participant is unconscious on Day 1 and receives the passive intervention, and thereafter becomes alert and cooperative on day 2, then he/she can receive the active intervention.
  Other Names: Cycle Ergometer; X Box 360 Kinect

SUMMARY:
Critically ill patients are often confined to bedrest, because of the nature of their illness. However, it has now been shown that prolonged bedrest and immobility, particularly in critically ill adults and children, can lead to serious outcomes such as muscle weakness and prolonged stay in the intensive care unit (ICU). Research in adults has demonstrated that preventing immobility and introducing exercise and rehabilitation in adult patients early during their ICU illness can prevent these serious outcomes, reduce the duration of hospital stay, and enhance their recovery after they leave the ICU. The purpose of our research is to investigate if early mobilization and rehabilitation can also be performed in critically ill children, and eventually evaluate this results in beneficial outcomes in these children, as it has been shown to be in adults. However, given that children are not the same as adults, but have varying abilities to understand and participate in activities when they are sick, the investigators first have to evaluate the most appropriate and safe ways of helping children "exercise" while they are in the ICU. This objective of this study is to evaluate if 2 methods of rehabilitation (a stationary bike and interactive video game) can be implemented in critically ill children. These methods have been used in hospitalized children and in critically ill adults. The investigators will evaluate if these methods are safe for critically ill children.

DETAILED DESCRIPTION:
In this prospective cohort pilot study, eligible critically ill children aged 3 to 17 years will receive in addition to their usual care, a passive and/or an active mobility intervention, depending on their level of consciousness or cognitive ability. The active intervention will consist of an interactive video game (X Box 360 Kinect), while a cycle ergometer will be used as the passive intervention. The mobility interventions will be applied for a minimum of 10 minutes on day 1, and 20 minutes on day 2. For unconscious patients, or eligible patients who cognitively impaired, the passive intervention will be applied. As soon as the patient is conscious and cooperative, the active intervention will be applied.

The primary outcomes of interest in this pilot study are feasibility (defined as the ability to screen and enroll patients, consent rate and protocol adherence). Secondary outcomes of interest include safety outcomes, clinical outcomes and patient and caregiver satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Anticipated PCCU stay of more than 24 hours.
2. Clinical stable children at PCCU
3. Informed consent and or assent where appropriate
4. Agreement of the most responsible PCCU physician
5. Age ≥ 3years to < 18 years

Exclusion Criteria:

1. Hemodynamic instability, defined as requiring escalation in vasoactive agents or volume resuscitation within the preceding 4 hours. (Patients who are on stable or weaning doses of vasoactive agents will be considered eligible).
2. Anticipated death and/ or withholding of life-sustaining therapies
3. The presence of a contraindication to mobilization- e.g. Suspected or actual evidence of cerebral edema or elevated ICP, unstable spinal cord injuries, musculoskeletal injuries/ fixed deformities in the lower limbs (for the use of cycle ergometer) or the upper limbs (for the use of interactive video-gaming)
4. Unstable airway (defined as impending respiratory failure and/or endotracheal intubation is anticipated within the next 4 hours).
5. Patients who are already mobilizing well/or at their baseline level of function

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Feasibility | 2 days
  The primary outcome of interest in this pilot study is feasibility. Feasibility is defined as follows:
  1. The ability to screen and enroll eligible patients - enrolment rate of at least 70% of those approached for consent (benchmark for PCCU trials)
  2. Time to application of acute rehabilitation intervention.
  3. Protocol adherence - a protocol violation rate of < 10%.

SECONDARY OUTCOMES:
Safety | Study period
  The proportion of patients with adverse events attributable to the rehabilitation intervention (e.g. cardiorespiratory events, tube dislodgement's).
Change in activity from baseline | From baseline to end of intervention
  Change in activity from baseline, during and following the intervention as measured by accelerometer, and patient
Caregiver/user perception of intervention | At end of study period
  Self-administered survey of caregiver and or user, to evaluate perceptions of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Karen Choong, MB, BCh, MSc, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada